CLINICAL TRIAL: NCT03553784
Title: Evaluating Process and Effectiveness of Low-intensity Group Cognitive Behavioural Therapy for Women With Gynaecological Cancer: The EPELIT Study
Brief Title: Low-Intensity CBT for Gynaecological Cancer Survivors
Acronym: EPELIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chester (Other)
Responsible Party: Principal Investigator, Nicholas J. Hulbert-Williams, Professor, University of Chester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 239518
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Gynecological Cancer
Keywords: Cancer; Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A pragmatic non-randomized controlled design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Group delivered Low Intensity Cognitive Behavioural Therapy (CBT).
  Interventions: Other: Group delivered Low Intensity Cognitive Behavioural Therapy
- Control Group (No Intervention): No intervention.

INTERVENTIONS:
Other: Group delivered Low Intensity Cognitive Behavioural Therapy — The intervention is group-delivered, low-intensity CBT similar to that used in IAPT (Improving Access to Psychological Therapies) Services in England. This intervention is already being offered as part of standard care at the Intervention site, and will not be altered by the study protocol, other than the requirement to complete a few more questionnaires. The intervention group meets weekly for eight weeks, and is facilitated by a clinical psychologist, a psychological well-being practitioner and a clinical nurse specialist from the medical oncology team. Content of the intervention is broad CBT, combining aspects of second-wave CBT, with elements of Narrative Therapy and ACT.
  Arms: Intervention Group

SUMMARY:
There are 21,500 gynaecological cancers diagnosed in the UK each year. These are often diagnosed later than common cancers, which is predictive of low survival and high psychological distress. There are few studies published which accurately map the profile of distress and supportive care needs in gynaecological cancer patients, nor which test psychological interventions to support this group.

This study will use a non-randomised controlled trial design to explore the potential benefits of taking part in a psychological intervention designed in this group of women. The intervention is group-delivered and runs for eight weeks. It is delivered by psychologists, psychological wellbeing practitioners, and cancer nurse specialists. The investigators will use validated self-report questionnaires to assess how helpful this intervention is at reducing distress and improving quality of life in the participants. This will be done in comparison with a treatment-as-usual control group recruited from a second clinical site. This second group of participants will not receive the psychological intervention, but they will complete the same assessments, at the same time points. To ensure participants are well supported, data collection in control control group participants will be done by telephone interview rather than self-report questionnaires. Both groups of participants will undertake a three-month follow-up assessment to check the longer-term effectiveness of the psychological intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be over the age of 16.
* Must have received a gynecological cancer diagnosis.
* Must have completed first line treatment within four months of the study start date (not restricted to any specific modality of treatment).
* Must be able to speak English.
* Must be able to provide consent.

Exclusion Criteria:

* Any patients that are unlikely to survive for the full five-month duration of the study.
* Any patient who does not have sufficient English language ability to complete data collection.
* Any patients who are notable to provide consent will not be included as this group would be unlikely to be able to complete data collection even if adjustments to the consent procedure were made.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | last 2 weeks
  A nine-item screening tool to assess symptoms of depression in the responding individual (Kroenke, Spitzer, & Williams, 2001). The PHQ-9 uses a four-point rating scale (ranging from 0 to 3) asking how often in the last two weeks participants have experienced symptoms pertaining to appetite, concentration, energy hopelessness, and suicidality. Higher scores indicate higher levels of distress. The PHQ-9 has been established as a valid and reliable measure of depression severity (Kroenke et al., 2001).
Generalized Anxiety Disorder (GAD-7) | last 2 weeks
  A seven-item screening tool to assess symptoms of anxiety in the responding individual (Spitzer, Kroenke, Williams, & Löwe, 2006). The GAD-7 uses a four-point rating scale (ranging from 0 to 3) asking how often in the last two weeks participants have experienced symptoms pertaining to feeling anxious, worried, difficulty relaxing, and irritability. Higher scores indicate higher distress. The GAD-7 has been established as an accurate measure of anxiety (Swinson, 2006).

SECONDARY OUTCOMES:
The Functional Assessment of Cancer Therapy-General (FACT-G) | last 7 days
  A 33-item screening tool to assess quality-of-life in patients receiving cancer treatment (Cella et al., 1993). The FACT-G uses a five-point rating scale (ranging from 0 to 4) asking how often in the last seven days patients have experienced difficulties in four dimensions of well-being: physical; social/family; emotional; functional. Higher scores indicate lower quality-of-life. The FACT-G is a well validated tool for measuring quality-of-life in cancer sample (Luckett et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Hulbert-Williams, PhD, Principal Investigator — University of Chester
Locations (1):
- Chester Research Unit for the Psychology of Health, Chester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised dataset will be prepared once our study is completed, primarily to ensure that access can be provided to journal editors and peer reviewers if requested through the publishing and dissemination process. We would consider requests to share this data with other research teams, provided that individual participants have consented to this .
  In releasing such data we will include self-report psychological measures, demographics as reported to the research team by the participant, and clinical data as extracted from patient records. We will not release information on hospital site, simply reporting that participants were recruited from anonymised UK hospitals. Thus, without access to how these match NHS records, it ought not to be possible to identify individuals from this dataset. This is carefully explained to participants in the study information sheets as an assurance of commitment to participant anonymity.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: We will make data available to others wishing to verify our analyses from the end of the study onward. We will impose a 24-month embargo after study end before releasing data for use for new analyses to other research teams.
Access Criteria: To be developed by our Study Steering Group nearer to the end of study completion

REFERENCES:
- [Derived] Hulbert-Williams NJ, Hulbert-Williams L, Flynn RJ, Pendrous R, MacDonald-Smith C, Mullard A, Swash B, Evans G, Price A. Evaluating process and effectiveness of a low-intensity CBT intervention for women with gynaecological cancer (the EPELIT Trial). AMRC Open Res. 2021 Mar 29;3:12. doi: 10.12688/amrcopenres.12971.1. eCollection 2021. PMID 38708072